CLINICAL TRIAL: NCT06278688
Title: Precision Probiotic Supplementation in Individuals With Mild Cognitive Impairment: a Randomized Controlled Trial
Brief Title: Precision Probiotic Supplementation in Individuals With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency); Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112R10438Y
Record Dates: First submitted 2023-11-13; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision probiotics (Experimental): The precision probiotics will be designed based on the results of probiotic signatures and consensus clustering described in the PRELIMINARY AND SUPPORTING Data section and available probiotics from GenMont Biotech Inc. (https://www.genmont.com.tw/)
  Interventions: Dietary Supplement: Precision probiotics
- Placebo (wait-list group) (Placebo Comparator): Placebo packets or capsules will be composed of maize starch only and be identical in appearance, weight, and smell. After completing trials, the Placebo group will be provided with a 6- month precision probiotic supplement.
  Interventions: Dietary Supplement: Precision probiotics

INTERVENTIONS:
Dietary Supplement: Precision probiotics — The precision probiotics will be designed based on the results of probiotic signatures and consensus clustering described in the PRELIMINARY AND SUPPORTING Data section and available probiotics from GenMont Biotech Inc. (https://www.genmont.com.tw/) The individual gut microbiota will determine the supplement and composition of probiotics.

SUMMARY:
The overarching goal of this randomized-controlled trial is to investigate the role and mechanism of the microbiota-gut-brain axis in MCI. The main questions it aims to answer are:

Aim 1: To investigate the association between gut microbiota, MCI and AD biomarkers. Investigators plan to compare gut microbiota profiles in a well-characterized cohort between individuals with MCI and cognitively normal adults using metagenomics sequencing data. Also, the relationship between gut microbiota and AD biomarkers, such as amyloid PET and plasma tau, will be explored in MCI and cognitively normal adults.

Aim 2: To determine the efficacy of precision probiotic supplementation on cognitive decline (primary outcome) and functional brain changes (secondary outcome) in individuals with MCI due to AD using a randomized, double-blind, placebo-controlled trial. Investigators plan to recruit 120 individuals with MCI due to AD, i.e., MCI with positive amyloid biomarkers. Participants will be randomized to a 12-month supplement of precision probiotics based on the individual gut probiotic profile or placebo. The primary outcome measure will be the changes in cognitive functions over 6 months (primary endpoint) and 12 months. The secondary outcome measure will be resting-state functional brain changes.

Aim 3: To investigate potential mediators underlying the effect of probiotic supplementation. The most apparent mediator will be a shift or changes in gut microbiota. Other potential mediators will be related to decreased lipopolysaccharide, proinflammatory cytokines such as tumor necrosis factor-alpha (TNF-α), interleukin (IL)-6 and IL-10, and increased brain- derived neurotrophic factor, short-chain fatty acid, etc.

DETAILED DESCRIPTION:
Given the rapidly aging trend worldwide and in Taiwan, the disease burden and economic impact of dementia on families, healthcare systems, and society are expected to increase unprecedentedly. It is estimated that interventions that could delay the clinical onset of dementia by a modest one year would significantly reduce the prevalence of dementia. Mild cognitive impairment (MCI) presents an early stage of cognitive impairment with a much higher risk of progression to dementia and a unique stage, potentially amenable to intervention, preventing further decline to dementia.

The microbiota-gut-brain axis is one of the most-studied gut-organ systems, and accumulating evidence shows gut microbiota might play a critical role in the pathogenesis of Alzheimer's disease (AD). However, the role of gut microbiota in the early stage of the AD spectrum, such as MCI, is unclear. Also, the effects of the probiotic supplements on cognition in patients with AD or MCI from several small randomized-controlled trials were inconsistent. Fixed regimens of probiotics were used in all these trials, and patients with MCI diagnosed by diverse research frameworks were included. As a result, the overarching goal of this proposal is to investigate the role and mechanism of the microbiota-gut-brain axis in MCI. Investigators will use data from a well-characterized cohort and a randomized controlled trial with a "precision" probiotic supplementation, i.e., a probiotic supplement based on individual gut probiotic profile, in a group of MCI due to AD, i.e., MCI with positive amyloid biomarkers.

ELIGIBILITY:
Inclusion criteria:

* 60 years old and above
* Diagnosis of MCI based on 2011 NIA-AA criteria
* Amyloid (+) measured by either amyloid PET imaging or CSF amyloid markers
* No dietary supplements, including other probiotics, yogurts with live, active cultures or supplements, and immune-enhancing supplements in the past three months (or wash-out period for three months for individuals taking supplements)
* No use of antibiotics, anti-inflammatory medications, gastrointestinal medicine within the past three months (or wash-out period for three months for individuals taking medications)
* Consenting to be randomly assigned intervention

Exclusion criteria:

* Currently undergoing cancer treatment.
* The anticipated life expectancy of less than six months.
* Suffering from severe mental disorders such as schizophrenia, bipolar disorder, or major depressive disorder.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The changes in attention | baseline, 3 months, 6 months, 12 months postintervention
  The primary outcome measure is the change in standardized scores (z-scores) for attention after 12 months. The average of the standardized scores of forward and backward digit Span subtest, digit symbol substitution subtests and symbol Searching subtest of the Wechsler Adult Intelligence Scale-III (WAIS-3) will represent the score for that domain, with higher scores indicating better performance.
The changes in memory | baseline, 3 months, 6 months, 12 months postintervention
  The primary outcome measure is the change in scores for the memory after 12 months. In the memory domain, the Logical Memory subset of the Wechsler Memory Scale (Hua et al., 1997) will be used, with higher scores indicating better performance.
The changes in executive function | baseline, 3 months, 6 months, 12 months postintervention
  The primary outcome measure is the change in standardized scores (z-scores) for executive function after 12 months. The average of the standardized scores of the color trails test, stroop color and word test, and verbal fluency test will represent the score for that domain, with higher scores indicating better performance.

SECONDARY OUTCOMES:
The changes in global cognition at the 12th month from baseline. | baseline, 6months, 12 months postintervention
  Mental State Examination measures global cognition and screening tools for cognitive impairment in older, community-dwelling, hospitalized, and institutionalized adults. The education adjusted cut-off was used to indicate impaired global cognition. It has been translated into Chinese for clinical use in Taiwan. It has a maximum score of 30 points, with higher scores indicating better global cognition.
The changes in brain imaging at the 12th month from baseline. | baseline, 6months, 12 months postintervention
  The brain Magnetic Resonance Imaging (MRI) will be performed on a 3-Tesla Magnetom Scanner in the Far-Eastern Memorial Hospital or the Cardinal Tien Hospital. The scanning protocol will consist of the following: whole-brain T1 magnetization-prepared rapid gradient-echo sequence, T2-weighted turbo spin-echo sequence, FLAIR pulse sequence, diffusion tensor imaging, and 6-min resting-state fMRI imaging using gradient-echo echo-planar imaging. During the resting-state fMRI, patients will be told to relax with closed eyes without concentrating on anything particular.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ling Chiu, Study Chair — Far Eastern Memorial Hospital

IPD SHARING:
Plan to Share IPD: Undecided